CLINICAL TRIAL: NCT07301489
Title: Akershus Cardiac Examination (ACE) 5 Study: Pragmatic Randomized Controlled Trial of Lung Cancer Screening Plus Program to Improve Cardiovascular Risk Profile and Health in Individuals With Heavy Smoking History
Brief Title: Akershus Cardiac Examination (ACE) 5 Study
Acronym: ACE5
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Helge Rørvik Røsjø, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: REK-ID: 870751; 24/10475 (Other: Division of Research and Innovation, Akershus University Hospital, Norway)
Record Dates: First submitted 2025-11-26; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Heavy Smokers; Lung Cancer Screening; Cardiovascular Risk Profile; Cardiovascular Disease Prevention
Keywords: Heavy smokers; Lung cancer screening; Cardiovascular risk profile; Cardiovascular disease prevention; Chronic coronary syndrome; Atherosclerotic cardiovascular disease; Non-contrast, non-cardiac chest CT-based screening; Nurse-led follow-up program
MeSH Terms: conditions — Atherosclerosis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Single-center, pragmatic randomized controlled trial of a non-pharmacological intervention.
  The investigators will perform visual four-group classification of coronary artery calcification in all participants from the TIDL Study. All ACE 5 Study participants will be invited to a baseline visit and 1-year follow-up visit. Participants will be randomized 1:1 to a hospital-based, nurse-led follow-up program (Lung Cancer Screening Plus Program) or standard of care after the participant has signed written informed consent.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung cancer screening plus (Experimental): Hospital-based, nurse-led follow-up
  Interventions: Other: Lung Cancer Screening Plus Program
- Standard of Care (Other): General practitioner-led follow-up
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Lung Cancer Screening Plus Program — In the intervention group, hospital-based, nurse-led follow-up will be tested, including risk stratification and risk factor intervention. Individuals normally meet a study nurse twice during 12-months of follow-up. If needed, this will be supplemented by meeting with a study physician. Individuals are informed to contact the hospital for all pharmacological prescriptions during the 12-month period.
  Arms: Lung cancer screening plus
Other: Standard of Care — In the control group, the General Practitioner will decide treatment and activities to reduce risk factors, which is the current model for follow-up of heavy smokers in Norway.
  Arms: Standard of Care

SUMMARY:
Individuals with extensive smoking history have 2- to 3-fold increased risk of dying prematurely compared to age- and gender-matched peers. Historical data indicate that 55% of heavy smokers will die from cardiovascular disease (CVD), while approximately 5% will die from lung cancer. Lung cancer screening programs are currently being implemented worldwide, but efforts to reduce also CVD are not included.

The research group behind the ACE 5 Study are affiliated with the study team behind the implementation study of lung cancer screening in Norway ("Tidlig oppdagelse av lungekreft [TIDL]"). The TIDL Study have performed non-contrast, non-cardiac chest CT-based screening for lung cancer in 1000 individuals. Prior studies have demonstrated that a visual four-group classification of coronary artery calcification using non-contrast, non-cardiac chest CT images provide an easily available, non-invasive surrogate index for subclinical and established chronic coronary syndrome. Accordingly, the 2024 European Society of Cardiology guidelines for chronic coronary syndrome promotes that opportunistic screening for atherosclerotic CVD (ASCVD) should be performed when non-contrast, non-cardiac chest CT images are available ("IIa recommendation"). The investigators will now invite TIDL participants for a second study, the Akershus Cardiac Examination (ACE) 5 Study, which will assess whether intervention also against ASCVD ("Lung Cancer Screening Plus Program") will improve cardiovascular risk profile and cardiovascular health in individuals with heavy smoking history.

The ACE 5 Study will be a separate study with separate protocol and consent as the ACE 5 Study will focus on the prevention of CVD in individuals with heavy smoking history as add-on to lung cancer screening. The ACE 5 Study will assess the combined effect of (1) non-contrast, non-cardiac chest CT images as basis for ASCVD detection, and (2) the value of a hospital-based, nurse-led follow-up program to improve cardiovascular risk profile and cardiovascular health in individuals with heavy smoking history. Whether a Lung Cancer Screening Plus Program can improve cardiovascular risk profile and indices of improved cardiovascular health compared to the current strategy/standard in individuals with heavy smoking history is currently not known. The primary endpoint relates to status for cardiovascular risk profile after 1-year follow-up, and the study will use pre-defined cutoffs for the different risk factors based on relevant European Society of Cardiology (ESC) Guidelines, especially the 2021 ESC guidelines for primary prevention and the 2024 ESC guidelines for chronic coronary syndrome.

DETAILED DESCRIPTION:
Background - The pathophysiology of chronic coronary syndrome

Myocardial infarction is the number 1 cause of death among smokers. An underlying framework related to this project is the potential to detect and treat atherosclerotic cardiovascular disease (ASCVD), which primarily manifests as coronary artery disease (CAD), prior to the development of symptoms and clinical events. This is important as CAD could be an unstable condition where acute occlusion of coronary arteries will lead to immediate myocardial necrosis, which is referred to as acute myocardial infarction. Smoking is a principal risk factor for atherosclerotic plaques and later symptomatic CAD. Myocardial infarction has significant mortality, both in the acute phase and later due to post-infarction heart failure mortality as well as recurrent myocardial infarction. As many as 1/5 of all patients having a myocardial infarction experience sudden cardiac death as their first symptom. Strategies that can detect CAD prior to events that leads to symptoms (subclinical disease) is therefore highly desirable.

Background - Lung Cancer Screening Programs and risk stratification for CVD

Lung cancer screening programs represent an excellent opportunity to screen high-risk individuals for ASCVD. Non-contrast, non-cardiac chest CT is the cornerstone of lung cancer screening and performed in all lung cancer screening participants. With these CT scans, the investigators can assess coronary artery calcification (CAC) with acceptable accuracy, either by using the four-group visual score or other method, like calculating Agatston score or ordinal visual scores. Moreover, as contrast agents are not required for the cardiac assessment and there is no need for ECG-triggering or cardiac specific protocols, the CT scans will not represent any risk to participant health or put additional strain on health services performing lung cancer screening. Radiation from current CT scans for lung cancer screening is 1.5-3 mSv, which is below the background radiation.

The clinical value of CACS by both Agatston, ordinal visual scores and the four-group visual score has been demonstrated in several studies, and the investigators believe that specific characteristics of our screening population will make assessing coronary artery calcification especially valuable for identifying subclinical CAD in the ACE 5 Study population. Assessment of CAC is also recommended by the National Lipid Association and the 2016 SCCT/STR guidelines for coronary artery calcium scoring of non-contrast noncardiac chest CT scans. One caveat of using coronary artery calcification to screen for subclinical CAD in the general population has been a very small number of individuals with CACS=0 that still experience cardiovascular events during follow-up. While CAC=0 is considered the one most important negative risk factor, a study of CAC in the lung cancer screening setting with non-contrast noncardiac chest CT scans show that up to 10% of the scans with CAC=0 experienced a major cardiac event. Hence, it is suggested that when CAC is assessed in noncardiac chest CT scans, CAC=0 should not always lead to delayed or avoidance of pharmacotherapies.

Traditional risk models like SCORE 2 also has limitations. Although excellent calibrated in the general population to identify high-risk individuals, SCORE 2 (and other models) cannot separate individual subjects in a group where all met the criteria of intermediate to high risk (>7.5% risk of cardiovascular event over 10-year follow-up). Hence, in our lung cancer screening population the inclusion criteria of age 60-79 years and 35 pack years of tobacco exposure in the TIDL Study will make most participants in the ACE 5 Study classified as intermediate to high risk for future cardiovascular event. Moreover, from epidemiological studies in the same age group, the investigators found 62% of middle-aged individuals to have a diagnosis of hypertension (defined according to prior, conservative criteria with blood pressure ≥140/90 mmHg) and mean total cholesterol was 5.5 mmol/L12. Accordingly, the investigators recognize that most participants in the ACE 5 Study will be classified as at least intermediate risk for CVD, and that no further separation is possible based on the SCORE 2 risk model.

Strategies to detect and reduce risk factors for ASCVD

Identifying subclinical CAD with the visual four-group classification will only reduce cardiovascular events if one is able to reduce risk factor profile in affected individuals. Several lifestyle and pharmacological interventions are efficient to reduce disease progression in subclinical CVD. Smoking is a principal risk factor and all participants in TIDL have been offered participation in a smoking cessation program. Smoking cessation will be follow-up also in the ACE 5 Study. Additional risk factors for ASCVD include hypertension, elevated atherogenic lipids, type 2 diabetes mellitus (T2DM), and physical inactivity.

The investigators will inform participants randomized to the standard-of-care group of the results from visual four-group classification of coronary artery calcification and the clinical examination. The investigators will provide this information to the physician of the participants randomized to standard care, given that this is approved by the participant. The investigators will include key information about guideline-directed medical goals, which is also the primary endpoint of the ACE 5 Study, in the letter to the participants and relevant physicians in the standard care group. In the control group, the General Practitioner (GP) will decide treatment and activities to reduce risk factors, which is the current model for follow-up of heavy smokers in Norway.

In contrast, for the intervention group the study will test hospital-based, nurse-led follow-up, including risk stratification and risk factor intervention. This model is a copy of the Swedish model for cardiovascular follow-up which is a 12-month hospital-based ("infarkt mottagning), nurse-led ("infarkt sjöterska") follow-up. In the Swedish model, individuals normally meet nurse x 2 and physician x 1 during 12-months of follow-up. In addition, individuals are informed to contact the hospital for all pharmacological prescriptions during the 12-month period. For all patients randomized to the Lung Cancer Screening Plus Program, the research team will perform an individual multidisciplinary assessment using the risk factors of each individual together with SCORE2 and coronary artery calcification to reach a recommendation for preventive measures aimed at lipid and blood sugar modifying therapy, antihypertensive therapy, smoking cessation, and increased physical activity. At every hospital visit, close monitoring of major prevention goals for guideline-directed medical therapy (GDMT) are checked. The nurse will contact the physician if GDMT goals are not met and therapy will be intensified. Health personnel also talk to patients/ participants about symptoms, side effects, and other questions that may affect treatment adherence.

The Swedish model has proven important to increase number of individuals with optimal GDMT, including reporting 1 year after myocardial infarction that 50% of smokers have stopped smoking, 77% have reached blood pressure target, and 60% have reached cholesterol target. In contrast, less than 30% of Norwegian patients have optimal GDMT after myocardial infarction. Still, whether the Swedish model for follow-up can be transferred also to a lung cancer screening program, and whether this model provides superior results to a strong GP-based health system, are currently not known.

Rationale for the Study

Individuals with extensive smoking history have 2- to 3-fold increased risk of dying prematurely compared to age- and gender-matched peers. Historical data indicate that 55% of heavy smokers will die from atherosclerotic cardiovascular disease (CVD), while approximately 5% will die from lung cancer. Lung cancer screening programs are currently being implemented worldwide, while no screening program has been developed for CVD. To utilize lung cancer screening programs as a basis for early detection of subclinical ASCVD in heavy smokers and to implement cost-efficient systems for risk reduction, should therefore be clinically relevant.

The research group behind the ACE 5 Study are affiliated with the study team behind the implementation study of lung cancer screening in Norway ("Tidlig oppdagelse av lungekreft [TIDL]"). Inclusion criteria for the TIDL Study include age 60-79 years and 35 pack years of tobacco exposure. The inclusion criteria will categorize most participants as at least intermediate risk for CVD during the next decade. As non-contrast, non-cardiac chest CT images, obtained during regular lung cancer screening, directly can assess atherosclerotic cardiovascular burden, it is hypothesized that additions to current lung cancer screening programs concomitantly will reduce CVD risk. In short, the ACE 5 Study will invite 1000 heavy smokers for baseline characterization, including blood sampling. After initial examination, calculation of SCORE 2 and visual four-group classification of CAC, the study will randomize (A) 50% of the participants to the intervention group with hospital-based, nurse-led follow-up and (B) 50% of the participants to the control group.

Study objectives

The TIDL Study has examinations of 1000 participants with non-contrast, non-cardiac chest CT and the ACE 5 Study should be able to include approximately 500 participants in each group. Only participants with complete follow-up data after 12 months are eligible for the primary endpoint, and an additional 5-10% drop out for the second visit is to be expected. The total number of participants in each group with complete data for the primary endpoint is expected to be around 450.

Primary endpoint

To determine whether a Lung Cancer Screening Plus Program in individuals with heavy smoking history improves cardiovascular risk profile, defined as reaching treatment goals or started new GDMT for smoking, lipid concentrations, blood pressure, and HbA1c, compared to the current strategy/standard care.

Study population The ACE 5 Study will enroll a maximum of 1000 participants meeting all inclusion criteria and no exclusion criteria. Only participants that have already consented to participate in the pilot implementation study for lung cancer screening in Norway ("Tidlig oppdagelse av lungekreft [TIDL]") are eligible for inclusion in the ACE 5 Study as these individuals have non-contrast, non-cardiac chest CT images available from the lung cancer screening study.

All patients will be thoroughly informed about all aspects of the study and the study team will collect informed, written consent from all study participants. Regardless of the time, at the request by the participant and not already included in a publication, all data collected in the study relating to the particular participant will be terminated.

There will be no restrictions to the diagnostic testing of our study participants, regardless of randomization status in the study. The decision of the patient to participate in the ACE 5 Study will not influence treatment that is offered to the patient at Akershus University Hospital and patients not participating in the study will receive current strategy/ standard care.

ELIGIBILITY:
Inclusion Criteria used for the lung cancer screening implementation study/ TIDL Study:

* Women and men
* Ages 60 to 79 years old (inclusive)
* A smoking history of at least 35 pack-years and 1) being a current smoker or a former smoker who quit less than 10 years prior or 2) having a PLCOm2012 model 6-year risk for lung cancer incidence over 2.6%.
* Willingness and ability to comply with scheduled visits, laboratory tests, and other trial procedures
* Written informed consent obtained prior to performing any protocol-related procedures
* The participant should be affiliated to a social security system

Exclusion Criteria used for the lung cancer screening implementation study/ TIDL Study:

* Recent abnormal pulmonary findings under work-up of standard care
* Having had chest CT <1 year before potential entry into the study
* Current or prior history of lung cancer, renal cancer, melanoma or breast cancer
* Inability to provide signed informed consent
* Insufficient understanding of the languages in which trial information is available
* Psychiatric or other disorders that are incompatible with compliance to the protocol requirements and follow-up
* Unable to be followed-up for at least 5-years
* Body weight >140 Kg because of difficulty of conducting the CT exam

Inclusion Criteria used for the ACE 5 Study:

* Participants from the TIDL Study with non-contrast, non-cardiac chest CT images available as part of the implementation lung cancer screening study
* Signed consent for cardiovascular add on-study and agree to protocol, including follow-up visit 1-year after the baseline examination

Exclusion Criteria used for the ACE 5 Study:

* Any surgical or medical condition, including short life-expectancy, based on medical records or clinical findings prior to randomization, that will impair the ability of the patient to participate in the study
* Patients unwilling or unable to comply with the protocol
* History of non-compliance to medical management and patients who are considered potentially unreliable, based on information obtained prior to randomization
* History or evidence of alcohol or drug abuse with the last 12 months, based on information obtained prior to randomization, that will influence study participation

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2041-04 (Estimated)

PRIMARY OUTCOMES:
Number of people reaching treatment goals or started new GDMT for smoking, lipid concentrations, blood pressure, and HbA1c | 12 months from the baseline visit
  To determine whether a Lung Cancer Screening Plus Program in individuals with heavy smoking history improves cardiovascular risk profile, defined as reaching treatment goals or started new GDMT for smoking, lipid concentrations, blood pressure, and HbA1c, compared to the current strategy/standard care.
  Treatment targets are defined as following:
  1. LDL cholesterol < 1.4 or started treatment with statin and/or ezetimibe after baseline visit
  2. Blood pressure <130/80 or started new antihypertensive therapy after baseline visit
  3. No smoking
  4. HbA1c < 52 mmol/L or started new antidiabetic therapy after baseline visit

SECONDARY OUTCOMES:
Number of people with lipid lowering treatment, antihypertensive treatment and antidiabetic treatment at 12 months | 12 months from the baseline visit
  To estimate change in lipid lowering treatment, antihypertensive treatment and antidiabetic treatment 12 months after the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Prevalence of smoking at 12 months post the baseline visit | 12 months from the baseline visit
  To estimate change in smoking prevalence at 12 months post the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Blood lipid concentrations at 12 months post the baseline visit | 12 months after the baseline visit
  To estimate change in blood lipid concentrations at 12 months post the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Blood pressure at 12 months post the baseline visit | 12 months after the baseline visit
  To estimate change in blood pressure at 12 months post the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
HbA1c concentrations at 12 months post the baseline visit | 12 months after the baseline visit
  To estimate change in HbA1c at 12 months post the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Rate of adherence to guideline directed medical therapy for ASCVD at 12 months post the baseline visit | 12 months after the baseline visit
  To estimate the difference in guideline directed medical therapy for ASCVD, as defined by international guidelines, at 12 months post the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Activity quotient at 12 months post the baseline visit | 12 months after the baseline visit
  To estimate change in self-reported physical activity at 12 months post the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history.
  An activity quotient will be calculated from participants' self-reported physical activity. They will be asked about frequency, duration, and intensity of exercise.
  Frequency of physical activity will be assessed by the question: "how often do you exercise" with the following response options: "never", "less than once a week", "once a week", "2-3 times a week", or "nearly every day".
  Those who reported engaging in physical activity at least once a week will be asked to assess their exertion level with three options: "exercising at a low intensity without becoming breathless", "exercising at a moderate intensity leading to breathlessness and sweating" or "engaging in vigorous exercise to near exhaustion".
  Duration of physical activity was assessed wit
Quality-of-life (EQ-5D-5L) at 12 months post the baseline visit | 12 months after the baseline visit
  To estimate change in quality-of-life (EQ-5D-5L) at 12 months post the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Glomerular filtration rate at 12 months post the baseline visit | 12 months after the baseline visit
  To estimate change in estimated glomerular filtration rate at 12 months post the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Time to the first event (either [1] any atherosclerotic cardiovascular event or intervention, or [2] non-cancer-related mortality) | Data will be reported at the 1 year follow-up, and at 5 years, 8 years, 10 years, 13 years, and 15 years for secondary endpoints.
  To determine whether a Lung Cancer Screening Plus Program in individuals with heavy smoking history reduces the time to the first event for either (1) any atherosclerotic cardiovascular event or intervention, or (2) non-cancer-related mortality, i.e. time to the combined endpoint, compared to the current strategy/ standard care
Time to non-cancer-related mortality | Data will be reported at the 1 year follow-up, and at 5 years, 8 years, 10 years, 13 years, and 15 years for secondary endpoints.
  To assess whether the Lung Cancer Screening Plus Program extends time to non-cancer-related mortality compared to current strategy/ standard care in individuals with heavy smoking history
Time to all-cause mortality | Data will be reported at the 1 year follow-up, and at 5 years, 8 years, 10 years, 13 years, and 15 years for secondary endpoints.
  To assess whether the Lung Cancer Screening Plus Program extends time to all-cause mortality compared to current strategy/ standard care in individuals with heavy smoking history
Time to any cardiovascular event or intervention | Data will be reported at the 1 year follow-up, and at 5 years, 8 years, 10 years, 13 years, and 15 years for secondary endpoints.
  To assess whether the Lung Cancer Screening Plus Program extends time to any cardiovascular event or intervention from the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Total number of any cardiovascular events or interventions | Data will be reported at the 1 year follow-up, and at 5 years, 8 years, 10 years, 13 years, and 15 years for secondary endpoints.
  To assess whether the Lung Cancer Screening Plus Program reduces the total number of any cardiovascular events or interventions from the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Total number of coronary events or interventions | Data will be reported at the 1 year follow-up, and at 5 years, 8 years, 10 years, 13 years, and 15 years for secondary endpoints.
  To assess whether the Lung Cancer Screening Plus Program reduces the total number of coronary events or interventions during follow-up for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Difference in total cost | Data will be reported at the 1 year follow-up, and at 5 years, 8 years, 10 years, 13 years, and 15 years for secondary endpoints.
  To estimate the difference in total cost from the baseline visit for participants in the Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history
Cost-utility | Data will be reported at the 1 year follow-up, and at 5 years, 8 years, 10 years, 13 years, and 15 years for secondary endpoints.
  To estimate cost-utility, i.e. cost per quality-adjusted life years gained, for the strategy with Lung Cancer Screening Plus Program compared to current strategy/ standard care in individuals with heavy smoking history

CONTACTS AND LOCATIONS:
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data (marked with study code) will be shared with national and international collaborators, e.g. for deep Phenotyping and Exploratory Endpoints.
Supporting Information: Study Protocol, SAP, Analytic Code
Access Criteria: Only de-identified data (marked with study code) will be shared with national and international collaborators.

REFERENCES:
- [Background] Garratt AM, Stavem K, Shaw JW, Rand K. EQ-5D-5L value set for Norway: a hybrid model using cTTO and DCE data. Qual Life Res. 2025 Feb;34(2):417-427. doi: 10.1007/s11136-024-03837-3. Epub 2024 Nov 20. PMID 39565555
- [Background] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710
- [Background] Sverre E, Peersen K, Perk J, Husebye E, Gullestad L, Dammen T, Otterstad JE, Munkhaugen J. Challenges in coronary heart disease prevention - experiences from a long-term follow-up study in Norway. Scand Cardiovasc J. 2021 Apr;55(2):73-81. doi: 10.1080/14017431.2020.1852308. Epub 2020 Dec 4. PMID 33274648
- [Background] Jernberg T, Attebring MF, Hambraeus K, Ivert T, James S, Jeppsson A, Lagerqvist B, Lindahl B, Stenestrand U, Wallentin L. The Swedish Web-system for enhancement and development of evidence-based care in heart disease evaluated according to recommended therapies (SWEDEHEART). Heart. 2010 Oct;96(20):1617-21. doi: 10.1136/hrt.2010.198804. Epub 2010 Aug 27. PMID 20801780
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Berge T, Lyngbakken MN, Ihle-Hansen H, Brynildsen J, Pervez MO, Aagaard EN, Vigen T, Kvisvik B, Christophersen IE, Steine K, Omland T, Smith P, Rosjo H, Tveit A. Prevalence of atrial fibrillation and cardiovascular risk factors in a 63-65 years old general population cohort: the Akershus Cardiac Examination (ACE) 1950 Study. BMJ Open. 2018 Aug 1;8(7):e021704. doi: 10.1136/bmjopen-2018-021704. PMID 30068617
- [Background] SCORE2 working group and ESC Cardiovascular risk collaboration. SCORE2 risk prediction algorithms: new models to estimate 10-year risk of cardiovascular disease in Europe. Eur Heart J. 2021 Jul 1;42(25):2439-2454. doi: 10.1093/eurheartj/ehab309. PMID 34120177
- [Background] Hecht HS, Cronin P, Blaha MJ, Budoff MJ, Kazerooni EA, Narula J, Yankelevitz D, Abbara S. 2016 SCCT/STR guidelines for coronary artery calcium scoring of noncontrast noncardiac chest CT scans: A report of the Society of Cardiovascular Computed Tomography and Society of Thoracic Radiology. J Cardiovasc Comput Tomogr. 2017 Jan-Feb;11(1):74-84. doi: 10.1016/j.jcct.2016.11.003. Epub 2016 Nov 10. PMID 27916431
- [Background] Orringer CE, Blaha MJ, Blankstein R, Budoff MJ, Goldberg RB, Gill EA, Maki KC, Mehta L, Jacobson TA. The National Lipid Association scientific statement on coronary artery calcium scoring to guide preventive strategies for ASCVD risk reduction. J Clin Lipidol. 2021 Jan-Feb;15(1):33-60. doi: 10.1016/j.jacl.2020.12.005. Epub 2020 Dec 11. PMID 33419719
- [Background] Greenland P, Bonow RO, Brundage BH, Budoff MJ, Eisenberg MJ, Grundy SM, Lauer MS, Post WS, Raggi P, Redberg RF, Rodgers GP, Shaw LJ, Taylor AJ, Weintraub WS; American College of Cardiology Foundation Clinical Expert Consensus Task Force (ACCF/AHA Writing Committee to Update the 2000 Expert Consensus Document on Electron Beam Computed Tomography); Society of Atherosclerosis Imaging and Prevention; Society of Cardiovascular Computed Tomography. ACCF/AHA 2007 clinical expert consensus document on coronary artery calcium scoring by computed tomography in global cardiovascular risk assessment and in evaluation of patients with chest pain: a report of the American College of Cardiology Foundation Clinical Expert Consensus Task Force (ACCF/AHA Writing Committee to Update the 2000 Expert Consensus Document on Electron Beam Computed Tomography) developed in collaboration with the Society of Atherosclerosis Imaging and Prevention and the Society of Cardiovascular Computed Tomography. J Am Coll Cardiol. 2007 Jan 23;49(3):378-402. doi: 10.1016/j.jacc.2006.10.001. No abstract available. PMID 17239724
- [Background] Xie X, Zhao Y, de Bock GH, de Jong PA, Mali WP, Oudkerk M, Vliegenthart R. Validation and prognosis of coronary artery calcium scoring in nontriggered thoracic computed tomography: systematic review and meta-analysis. Circ Cardiovasc Imaging. 2013 Jul;6(4):514-21. doi: 10.1161/CIRCIMAGING.113.000092. Epub 2013 Jun 11. PMID 23756678
- [Background] Handy CE, Quispe R, Pinto X, Blaha MJ, Blumenthal RS, Michos ED, Lima JAC, Guallar E, Ryu S, Cho J, Kaye JA, Comin-Colet J, Corbella X, Cainzos-Achirica M. Synergistic Opportunities in the Interplay Between Cancer Screening and Cardiovascular Disease Risk Assessment: Together We Are Stronger. Circulation. 2018 Aug 14;138(7):727-734. doi: 10.1161/CIRCULATIONAHA.118.035516. PMID 30359131
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Carlhed R, Bojestig M, Wallentin L, Lindstrom G, Peterson A, Aberg C, Lindahl B; QUICC study group. Improved adherence to Swedish national guidelines for acute myocardial infarction: the Quality Improvement in Coronary Care (QUICC) study. Am Heart J. 2006 Dec;152(6):1175-81. doi: 10.1016/j.ahj.2006.07.028. PMID 17161072
- [Background] Chiles C, Duan F, Gladish GW, Ravenel JG, Baginski SG, Snyder BS, DeMello S, Desjardins SS, Munden RF; NLST Study Team. Association of Coronary Artery Calcification and Mortality in the National Lung Screening Trial: A Comparison of Three Scoring Methods. Radiology. 2015 Jul;276(1):82-90. doi: 10.1148/radiol.15142062. Epub 2015 Mar 9. PMID 25759972
- [Background] Benowitz NL. Nicotine addiction. N Engl J Med. 2010 Jun 17;362(24):2295-303. doi: 10.1056/NEJMra0809890. No abstract available. PMID 20554984
- [Background] Abrams J. Clinical practice. Chronic stable angina. N Engl J Med. 2005 Jun 16;352(24):2524-33. doi: 10.1056/NEJMcp042317. No abstract available. PMID 15958808
- [Background] Doll R, Peto R, Boreham J, Sutherland I. Mortality in relation to smoking: 50 years' observations on male British doctors. BMJ. 2004 Jun 26;328(7455):1519. doi: 10.1136/bmj.38142.554479.AE. Epub 2004 Jun 22. PMID 15213107